CLINICAL TRIAL: NCT05916937
Title: Extending Omalizumab Treatment Intervals in Patients With Chronic Spontaneous Urticaria (EXOTIC Trial): a Multicentre, Randomized, Open-label, Non-inferiority Trial
Brief Title: Extending Omalizumab Treatment Intervals in Patients With Chronic Spontaneous Urticaria
Acronym: EXOTIC
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Simon Francis Thomsen (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor-Investigator, Simon Francis Thomsen, DM, PhD, DMSc, Bispebjerg Hospital
Organization: Bispebjerg Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: p-2023-14337
Record Dates: First submitted 2023-06-06; First posted 2023-06-23 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2024-10

CONDITIONS: Chronic Spontaneous Urticaria; Chronic Urticaria, Idiopathic
MeSH Terms: conditions — Chronic Urticaria | interventions — Omalizumab

STUDY DESIGN:
Intervention Model Description: Multicenter, randomized, open-label, non-inferiority trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- omalizumab 300 mg every six weeks (Active Comparator): 20 subjects are randomized to receive omalizumab 300 mg every six weeks from week 12 to week 36.
  Interventions: Drug: omalizumab 300 mg every six weeks
- omalizumab 300 mg every four weeks (Active Comparator): 20 subjects are randomized to receive omalizumab 300 mg every four weeks from week 12 to week 36.
  Interventions: Drug: omalizumab 300 mg every four weeks

INTERVENTIONS:
Drug: omalizumab 300 mg every four weeks — Continue standard treatment with omalizumab 300 mg every four weeks from week 12 to week 36.
  Both arms are treated with omalizumab 300 mg from week 0 to week 12.
  Other Names: Standard treatment
  Arms: omalizumab 300 mg every four weeks
Drug: omalizumab 300 mg every six weeks — Treatment in an extended interval of omalizumab 300 mg every six weeks from week 12 to week 36.
  Both arms are treated with omalizumab 300 mg from week 0 to week 12.
  Other Names: Extended treatment
  Arms: omalizumab 300 mg every six weeks

SUMMARY:
This study is a multicentre, randomized, open-label, non-inferiority clinical trial.

The purpose and aim of this study is to investigate if patients with well controlled (UCT score score ≥ 12) chronic spontaneous urticaria (CSU) on omalizumab 300 mg every four weeks can extend treatment intervals and maintain disease control.

DETAILED DESCRIPTION:
Newly referred patients with CSU who are well-treated (UCT score ≥ 12) 12 weeks after initiating standard treatment with omalizumab 300 mg every four weeks, are randomized into two treatment arms.The first arm will continue standard treatment with omalizumab 300 mg every four weeks for 24 weeks. The second arm will receive treatment in an extended interval of omalizumab 300 mg every six weeks for 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of CSU according to the EAACI/GA2LEN/EDF/WAO guidelines.
* Age ≥ 18 years.
* Omalizumab-naïve prior to initiating treatment with omalizumab.
* Background treatment with four antihistamines daily.
* Candidate for omalizumab treatment according to Danish guidelines.

Exclusion Criteria:

* Pregnant or breastfeeding women.
* Planned pregnancy within the next 6 months.
* Weight ≥ 100 kilograms.
* Presence of any other active skin disease or condition that may interfere with the assessment of CSU, such as atopic dermatitis, bullous pemphigoid, senile pruritus, or psoriasis.
* Use of immunosuppressive drugs, such as prednisolone, azathioprine, methotrexate, or cyclosporine.
* Predominantly experience symptoms from chronic inducible urticaria (CIndU).
* Inability to complete study or comply with study procedures.

Patients with a positive basophil histamine release assay (BHRA) are not eligible for the study. Patients may therefore be withdrawn from the trial after enrolment, if they are found to have a positive BHRA test in the initial blood work.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-01-12 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Absolute difference in average Urticaria Control Test (UCT) score at week 36 | Through study completion, an average of 36 weeks
  The Urticaria Control Test (UCT) is a retrospective questionnaire that gathers information regarding the past 4 weeks. It consists of four questions, each with four possible answer options. A score ranging from 0 to 4 is assigned to each answer option. Consequently, the UCT score ranges from 0 to 16, with higher scores indicating lower control of the disease. A UCT score of 12 or higher suggests well-controlled urticaria, while a score of 16 indicates complete control.

SECONDARY OUTCOMES:
Absolute difference in average Urticaria Control Test (UCT) score at week 24 | Through study completion, an average of 36 weeks
  The Urticaria Control Test (UCT) is a retrospective questionnaire that gathers information regarding the past 4 weeks. It consists of four questions, each with four possible answer options. A score ranging from 0 to 4 is assigned to each answer option. Consequently, the UCT score ranges from 0 to 16, with higher scores indicating lower control of the disease. A UCT score of 12 or higher suggests well-controlled urticaria, while a score of 16 indicates complete control.
Proportion of well-controlled patients (UCT score ≥ 12) at week 24 and 36 | Through study completion, an average of 36 weeks
  The Urticaria Control Test (UCT) is a retrospective questionnaire that gathers information regarding the past 4 weeks. It consists of four questions, each with four possible answer options. A score ranging from 0 to 4 is assigned to each answer option. Consequently, the UCT score ranges from 0 to 16, with higher scores indicating lower control of the disease. A UCT score of 12 or higher suggests well-controlled urticaria, while a score of 16 indicates complete control.
Proportion of completely controlled patients (UCT score = 16) at week 24 and 36 | Through study completion, an average of 36 weeks
  The Urticaria Control Test (UCT) is a retrospective questionnaire that gathers information regarding the past 4 weeks. It consists of four questions, each with four possible answer options. A score ranging from 0 to 4 is assigned to each answer option. Consequently, the UCT score ranges from 0 to 16, with higher scores indicating lower control of the disease. A UCT score of 12 or higher suggests well-controlled urticaria, while a score of 16 indicates complete control.
Difference in absolute UCT score measured as area under the curve (AUC) | Through study completion, an average of 36 weeks
  The Urticaria Control Test (UCT) is a retrospective questionnaire that gathers information regarding the past 4 weeks. It consists of four questions, each with four possible answer options. A score ranging from 0 to 4 is assigned to each answer option. Consequently, the UCT score ranges from 0 to 16, with higher scores indicating lower control of the disease. A UCT score of 12 or higher suggests well-controlled urticaria, while a score of 16 indicates complete control.
Absolute difference in average weekly urticaria activity score (UAS7) at week 24 and 36 | Through study completion, an average of 36 weeks
  The Urticaria Activity Score (UAS) is a score recorded in a diary that assesses the severity of wheals and intensity of pruritus experienced within a 24-hour period. The total UAS score can range from 0 to 6. The UAS7 is calculated by summing the daily UAS scores over the past week. The UAS7 score ranges from 0 to 42, with higher scores indicating greater disease activity. A UAS7 score of less than 7 suggests well-controlled urticaria, while a score of 0 indicates complete control.
Proportion of well-controlled patients (UAS7 score < 7) at week 24 and 36 | Through study completion, an average of 36 weeks
  The Urticaria Activity Score (UAS) is a score recorded in a diary that assesses the severity of wheals and intensity of pruritus experienced within a 24-hour period. The total UAS score can range from 0 to 6. The UAS7 is calculated by summing the daily UAS scores over the past week. The UAS7 score ranges from 0 to 42, with higher scores indicating greater disease activity. A UAS7 score of less than 7 suggests well-controlled urticaria, while a score of 0 indicates complete control.
Proportion of completely controlled patients (UAS7 score = 0) at week 24 and 36 | Through study completion, an average of 36 weeks
  The Urticaria Activity Score (UAS) is a score recorded in a diary that assesses the severity of wheals and intensity of pruritus experienced within a 24-hour period. The total UAS score can range from 0 to 6. The UAS7 is calculated by summing the daily UAS scores over the past week. The UAS7 score ranges from 0 to 42, with higher scores indicating greater disease activity. A UAS7 score of less than 7 suggests well-controlled urticaria, while a score of 0 indicates complete control.
Differences in average Chronic Urticaria Quality of Life (CU-QoL) at week 24 and 36 | Through study completion, an average of 36 weeks
  The Chronic Urticaria Quality of Life Questionnaire (Cu-QoL) is a retrospective questionnaire that gathers information regarding the past 2 weeks. The Cu-QoL consists of 23 questions, each scored on a scale from 1 (indicating no complaints) to 5 (indicating many complaints). Higher scores on the Cu-QoL reflect a lower quality of life.
Differences in average dermatology life quality index (DLQI) at week 24 and 36 | Through study completion, an average of 36 weeks
  The Dermatology Life Quality Index (DLQI) is a validated, self-administered questionnaire consisting of 10 items. It measures the impact of skin disease on patients' quality of life based on their recall of experiences over the past week. The questionnaire covers various domains, including symptoms, feelings, daily activities, social interactions, leisure activities, work or studying, personal relationships, and treatment. Each question is scored on a scale of 0 to 3, resulting in a total score range from 0 (indicating no impact of skin disease on quality of life) to 30 (indicating the maximum impact on quality of life).
Proportion of patients in the two treatment arms who experience flares | Through study completion, an average of 36 weeks
  Flares refer to the exacerbation of symptoms that prompt patients to reach out to their healthcare provider and/or request intensified treatment.
Adverse event (AEs) and serious advese events (SAEs) | Through study completion, an average of 36 weeks
  Adverse events (AEs) encompass any unfavorable and/or unintended signs, incidents, symptoms, or diseases associated with omalizumab. This also includes laboratory results falling outside the reference range, although only laboratory results deemed clinically relevant will be examined. Any AEs occurring from the first administration of the trial medication until 8 days after the last administration of the trial medicine will be documented. Serious adverse events (SAEs) are defined as AEs or adverse reactions that lead to death, are life-threatening, require hospitalization or prolongation of existing hospitalization, result in persistent or significant disability or incapacity, or involve a congenital anomaly or birth defect.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Dermatology, Bispebjerg Hospital, Copenhagen, Copenhagen N, Denmark

IPD SHARING:
Plan to Share IPD: No
Due to Danish data protection laws, data sharing is not planned. However, data can be made available upon reasonable request, in compliance with Danish legislation.

REFERENCES:
- [Derived] Zhang DG, Sorensen JA, Ghazanfar MN, Ali Z, Vestergaard C, Thyssen J, Egeberg A, Thomsen SF. EXtending Omalizumab Treatment Intervals in patients with Chronic spontaneous urticaria (EXOTIC): protocol of a multicentre, randomised, open-label, non-inferiority trial. BMJ Open. 2025 Jan 6;15(1):e084987. doi: 10.1136/bmjopen-2024-084987. PMID 39762098